CLINICAL TRIAL: NCT07128394
Title: Exogenous Luteinizing Hormone Supplementation to Improve Embryo Quality in Patients With Excessive LH Suppression During a Long GnRH-Agonist Protocol: A Randomized Controlled Trial
Brief Title: Extra Luteinizing Hormone Improve Embryo Quality in IVF Patients With Low LH During Long GnRH-Agonist Treatment
Acronym: ELH-IVF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ-ELH-2025; BJHPA-2023-SZHYXZHQN-006 (Other: Beijing Health Sponsoring Organization)
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Infertility, Female; Luteinizing Hormone (LH)
Keywords: Luteinizing Hormone; Long GnRH Agonist Protocol; Excessive LH Suppression; Controlled Ovarian Stimulation; In Vitro Fertilization; Embryo Quality
MeSH Terms: conditions — Infertility, Female | interventions — Luteinizing Hormone; Luteinizing Hormone, beta Subunit; Glycoprotein Hormones, alpha Subunit; follitropin alfa; Gonadotropin-Releasing Hormone; Triptorelin Pamoate

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either the intervention group receiving exogenous luteinizing hormone (LH) supplementation in addition to the standard long GnRH agonist protocol, or the control group receiving the standard long GnRH agonist protocol without LH supplementation. Both groups will undergo controlled ovarian stimulation and in vitro fertilization (IVF) according to the study protocol.
Masking Description: Not applicable. This is an open-label trial in which both participants and investigators are aware of the assigned interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant LH Supplementation Group (Experimental): Participants receive controlled ovarian hyperstimulation (COH) using a long-acting GnRH agonist (triptorelin 3.75 mg) for pituitary downregulation, followed by recombinant FSH (rFSH) combined with recombinant LH (rLH) at a ratio of 2:1 starting on stimulation day. rLH administration continues throughout the stimulation phase, with gonadotropin doses adjusted based on follicular growth and hormone monitoring. Trigger is given when 2-3 leading follicles reach ≥18 mm, followed by oocyte retrieval, IVF/ICSI, and embryo quality assessment.
  Interventions: Drug: Recombinant Luteinizing Hormone (rLH); Drug: Recombinant Follicle-Stimulating Hormone (rFSH); Drug: Gonadotropin-Releasing Hormone Agonist (GnRH-a)
- Conventional rFSH-Only Group (Active Comparator): Participants receive the same long-acting GnRH agonist downregulation and rFSH stimulation protocol as the experimental arm, but without rLH supplementation. Only rFSH is used during COH, with dose adjustments according to follicular development and hormone levels. Trigger, oocyte retrieval, IVF/ICSI, and embryo assessment follow the same procedures as in the experimental arm.
  Interventions: Drug: Recombinant Follicle-Stimulating Hormone (rFSH); Drug: Gonadotropin-Releasing Hormone Agonist (GnRH-a)

INTERVENTIONS:
Drug: Recombinant Luteinizing Hormone (rLH) — Recombinant LH administered subcutaneously in combination with recombinant FSH (rFSH) at a ratio of 2:1 starting on stimulation day, continued throughout controlled ovarian hyperstimulation. Dosage adjusted according to follicular growth and serum hormone levels.
  Other Names: lutropin alfa; Luveris
  Arms: Recombinant LH Supplementation Group
Drug: Recombinant Follicle-Stimulating Hormone (rFSH) — Recombinant FSH administered subcutaneously for controlled ovarian hyperstimulation after pituitary downregulation with a long-acting GnRH agonist. Dosage adjusted based on follicular development and hormone monitoring.
  Other Names: follitropin alfa; Gonal-F
Drug: Gonadotropin-Releasing Hormone Agonist (GnRH-a) — Long-acting GnRH agonist (3.75 mg) administered subcutaneously on menstrual cycle day 2-4 for pituitary downregulation before controlled ovarian hyperstimulation.
  Other Names: triptorelin; Diphereline

SUMMARY:
This randomized controlled trial aims to evaluate whether supplementation with exogenous luteinizing hormone (LH) can improve embryo quality in patients undergoing in vitro fertilization (IVF) with a long gonadotropin-releasing hormone agonist (GnRH-a) protocol who have excessive suppression of LH. Eligible participants will be randomly assigned to receive either exogenous LH supplementation or standard care. The primary outcome is embryo quality, and secondary outcomes include pregnancy rates and safety assessments. The study is conducted at Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University.

DETAILED DESCRIPTION:
Excessive suppression of luteinizing hormone (LH) during ovarian stimulation with a long gonadotropin-releasing hormone agonist (GnRH-a) protocol has been associated with suboptimal follicular development, impaired oocyte maturation, and reduced embryo quality. LH plays a critical role in the final stages of folliculogenesis, steroidogenesis, and ovulation, and its deficiency during controlled ovarian hyperstimulation may adversely affect the developmental competence of oocytes.

This randomized controlled trial is designed to evaluate whether supplementation with exogenous LH can improve embryo quality in patients undergoing in vitro fertilization (IVF) with excessive LH suppression during a long GnRH-a protocol. Eligible participants are women meeting predefined hormonal suppression criteria prior to or during stimulation. Participants will be randomly assigned to receive either exogenous LH supplementation in addition to standard ovarian stimulation or standard care without LH supplementation.

The primary endpoint is the proportion of high-quality embryos obtained per cycle. Secondary endpoints include clinical pregnancy rate, implantation rate, live birth rate, and safety outcomes such as incidence of ovarian hyperstimulation syndrome (OHSS) and adverse events.

The study aims to provide high-quality evidence to guide the optimal management of patients with profound LH suppression during controlled ovarian stimulation. Findings from this trial may contribute to refining stimulation protocols and improving reproductive outcomes in assisted reproductive technology (ART).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 to 37 years (inclusive). Diagnosed with infertility and undergoing in vitro fertilization/intracytoplasmic sperm injection (IVF/ICSI) treatment using the long-acting GnRH agonist protocol.

Serum luteinizing hormone (LH) level <0.5 U/L after pituitary downregulation. Normal uterine cavity as confirmed by hysteroscopy, sonohysterography, or hysterosalpingography within 6 months.

Written informed consent provided prior to participation.

Exclusion Criteria:

* Polycystic ovary syndrome (PCOS). History of recurrent implantation failure (RIF). Presence of endometriosis or adenomyosis. History of ovarian surgery. Ovarian cysts ≥3 cm or with suspected malignancy. Poor ovarian reserve (antral follicle count <5, anti-Müllerian hormone <1.1 ng/mL, or baseline FSH >10 IU/L).

Chromosomal abnormalities in either partner. Systemic diseases such as uncontrolled hypertension, diabetes, thyroid disorders, or autoimmune diseases.

Contraindications to ovarian stimulation medications or pregnancy.

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility is limited to biological females of reproductive age due to the study's focus on ovarian stimulation and embryo quality in IVF/ICSI cycles.
Enrollment: 590 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of cycles with no usable embryos | 7 days after oocyte retrieval
  The number of IVF/ICSI cycles with no transferable embryos divided by the total number of oocyte retrieval cycles, evaluated based on embryo morphology and grading on Day 3 or Day 5-6 after fertilization.

SECONDARY OUTCOMES:
Number of high-quality Day 3 embryos | 7 days after oocyte retrieval
  Count of embryos meeting morphological criteria for high quality on Day 3 after fertilization, as determined by standard embryology scoring.
Total gonadotropin dose used | At the end of ovarian stimulation (average 8-12 days)
  Cumulative dose (IU) of gonadotropins administered from stimulation start to trigger day.
Duration of gonadotropin stimulation | At the end of ovarian stimulation (average 8-12 days)
  Number of days from gonadotropin initiation to trigger day.
Number of oocytes retrieved | At oocyte retrieval (36-38 hours after trigger)
  Total number of oocytes collected during transvaginal ultrasound-guided oocyte retrieval.
Clinical pregnancy rate | 30 days after embryo transfer
  Proportion of embryo transfer cycles resulting in at least one intrauterine gestational sac with fetal heartbeat, confirmed by transvaginal ultrasound.
Early miscarriage rate | Within 12 weeks of gestation
  Proportion of clinical pregnancies ending in miscarriage before 12 completed weeks of gestation.
Live birth rate | At delivery (up to 1 year after embryo transfer)
  Proportion of embryo transfer cycles resulting in the delivery of at least one live-born infant.

CONTACTS AND LOCATIONS:
Overall Officials: 慧 Jiang, PhD, Principal Investigator — Nanjing Drum Tower Hospital: Nanjing University Medical School Affiliated Nanjing Drum Tower Hospital
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to concerns regarding patient privacy, confidentiality, and compliance with local regulations.

REFERENCES:
- [Background] Yazici Yilmaz F, Gorkemli H, Colakoglu MC, Aktan M, Gezginc K. The evaluation of recombinant LH supplementation in patients with suboptimal response to recombinant FSH undergoing IVF treatment with GnRH agonist down-regulation. Gynecol Endocrinol. 2015 Feb;31(2):141-4. doi: 10.3109/09513590.2014.965675. Epub 2014 Sep 19. PMID 25237892
- [Background] Tesarik J, Mendoza C. Effects of exogenous LH administration during ovarian stimulation of pituitary down-regulated young oocyte donors on oocyte yield and developmental competence. Hum Reprod. 2002 Dec;17(12):3129-37. doi: 10.1093/humrep/17.12.3129. PMID 12456612
- [Background] Wu KK, Papp AC, Manner CE, Hall ER. Interaction between lymphocytes and platelets in the synthesis of prostacyclin. J Clin Invest. 1987 Jun;79(6):1601-6. doi: 10.1172/JCI112995. PMID 3108319
- [Background] Kan O, Simsir C, Atabekoglu CS, Sonmezer M. The impact of adding hp-hMG in r-FSH started GnRH antagonist cycles on ART outcome. Gynecol Endocrinol. 2019 Oct;35(10):869-872. doi: 10.1080/09513590.2019.1600667. Epub 2019 Apr 11. PMID 30973022
- [Background] Propst AM, Hill MJ, Bates GW, Palumbo M, Van Horne AK, Retzloff MG. Low-dose human chorionic gonadotropin may improve in vitro fertilization cycle outcomes in patients with low luteinizing hormone levels after gonadotropin-releasing hormone antagonist administration. Fertil Steril. 2011 Oct;96(4):898-904. doi: 10.1016/j.fertnstert.2011.06.069. Epub 2011 Aug 11. PMID 21839437
- [Background] Tayyar AT, Kahraman S. Comparison between cycles of the same patients when using recombinant luteinizing hormone + recombinant follicle stimulating hormone (rFSH), human menopausal gonadotropin + rFSH and rFSH only. Arch Med Sci. 2019 May;15(3):673-679. doi: 10.5114/aoms.2017.72408. Epub 2018 Jan 8. PMID 31110533
- [Background] Fleming R, Rehka P, Deshpande N, Jamieson ME, Yates RW, Lyall H. Suppression of LH during ovarian stimulation: effects differ in cycles stimulated with purified urinary FSH and recombinant FSH. Hum Reprod. 2000 Jul;15(7):1440-5. doi: 10.1093/humrep/15.7.1440. PMID 10875848
- [Background] Westergaard LG, Laursen SB, Andersen CY. Increased risk of early pregnancy loss by profound suppression of luteinizing hormone during ovarian stimulation in normogonadotrophic women undergoing assisted reproduction. Hum Reprod. 2000 May;15(5):1003-8. doi: 10.1093/humrep/15.5.1003. PMID 10783342
- [Background] Alviggi C, Clarizia R, Mollo A, Ranieri A, De Placido G. Outlook: who needs LH in ovarian stimulation? Reprod Biomed Online. 2006 May;12(5):599-607. doi: 10.1016/s1472-6483(10)61186-8. PMID 16790105
- [Background] Li F, Ye T, Kong H, Li J, Hu L, Jin H, Su Y, Li G. Efficacies of different ovarian hyperstimulation protocols in poor ovarian responders classified by the POSEIDON criteria. Aging (Albany NY). 2020 May 29;12(10):9354-9364. doi: 10.18632/aging.103210. Epub 2020 May 29. PMID 32470947